CLINICAL TRIAL: NCT06546189
Title: Oral Lactobacillus Supplementation as Treatment for Overactive Bladder Syndrome: A Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marianne Koch, Priv.-Doz.Dr.med.univ., PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1917/2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): OMNi BiOTiC® 41167 sachet diluded in a glass of water twice daily oral intake for 6 months
  Interventions: Dietary Supplement: OMNi BiOTiC® 41167
- 2 (Placebo Comparator): Placebo sachet diluted in a glass of water twice daily oral intake for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OMNi BiOTiC® 41167 — The product "OMNi BiOTiC® 41167" contains lactobacillus strains
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
Background: Overactive bladder describes a syndrome characterized by frequent urges to urinate and increased urination with or without nocturia and with or without urinary incontinence. Overactive bladder affects approximately 13% of older women and thus represents a condition with high prevalence. Affected women report significant limitations in daily life, as well as social isolation. Despite the high occurrence of this condition, therapeutic options are limited, partly because the etiology of this condition is not fully understood. Increasingly, studies suggest an imbalance in the urogenital microbiome as a possible cause of the development of the condition. Therefore, the aim of this study is to test, whether the oral administration of a lactobacillus preparation can lead to a reduction in symptoms.

Design: Randomized controlled study

Methods: Intake of OMNi BiOTiC® 41167 or placebo twice daily for 6 months; swabs (vaginal and urethral) and urine samples from a single-use catheter for microbiome determination at 0, 3, and 7 months.

Outcome: Reduction of subjective symptoms (yes/no) after 3 and 7 months; reduction of Overactive Bladder Symptom Score after 3 and 7 months; change in the urogenital microbiome after 3 and 7 months (comparison of intervention vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of overactive bladder syndrome or mixed urinary incontinence with predominance of overactive bladder symptoms

Exclusion Criteria:

* under age 18
* neurogenic overactive bladder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
symptom reduction | 6 months
  yes/no
ICIQ-OAB symptom score reduction | 6 months

SECONDARY OUTCOMES:
change in vaginal/urethral/bladder microbiom | 3 months and 6 months
  between groups and within one participant

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided